CLINICAL TRIAL: NCT02301351
Title: Effects of Implicit Messaging by Cigarette Pack Color on Smoking Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Strasser, Research Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 819610; P50CA179546 (NIH)
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Cigarette Smoking Behavior
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Graphic Warning Label (Other): Days 5-50: Participants will receive cigarette packs as per the study randomization schema (e.g. three15-day periods of red, gold, and plain packs; order counterbalanced within subject) with FDA-approved graphic warning labels.
  Interventions: Other: Graphic Warning Label
- Text Warning Label (Other): Days 5-50: Participants will receive cigarette packs as per the study randomization schema (e.g. three15-day periods of red, gold, and plain packs; order counterbalanced within subject) with standard text warning labels.
  Interventions: Other: Text Warning Label

INTERVENTIONS:
Other: Graphic Warning Label — All packs provided will include FDA-approved graphic warning labels
  Arms: Graphic Warning Label
Other: Text Warning Label — All packs provided will include standard text warning labels
  Arms: Text Warning Label

SUMMARY:
The purpose of this study is to examine the effect of changes in cigarette package color and warning label features on smoking behaviors and beliefs about cigarette risks.

DETAILED DESCRIPTION:
This project will recruit 360, current daily Marlboro, non-menthol, red (n=180) or gold (n=180) cigarette smokers to a 50-day protocol using a randomized factorial design with two factors: (1) cigarette pack color manipulation (within subject: red, gold, plain packaging) and (2) warning label manipulation (between subject: graphic vs. standard text). The randomization will be stratified by own brand cigarette. To evaluate effects of changes in cigarette package coloring, participants will smoke commercially available cigarettes that may or may not be similar to their preferred brand of cigarettes throughout the study, but in different colored packages during three 15-day study periods (i.e., one period will be Marlboro plain (tan-olive) packs, one will be Marlboro gold packs and one will be Marlboro red packs; order counterbalanced). Participants will visit the Center every 5 days to complete assessments (11 total sessions).

ELIGIBILITY:
Inclusion Criteria:

* Male and female smokers who are between 21 and 60 years of age and self-report smoking at least 5 cigarettes per day for at least the past 12 months.
* Smokers of primarily non-menthol, Marlboro red or gold type cigarettes.
* Not using any forms of nicotine other than cigarettes.
* Not currently undergoing smoking cessation treatment or tying to quit.
* Able to communicate fluently in English (speaking, writing, and reading).
* Plan to remain in the area over the duration of the trial.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Exclusion Criteria:

Smoking Behavior.

* Use of any nicotine products other than cigarettes.
* Enrollment or plans to enroll in a smoking cessation program over the duration of the trial.
* Provide a Carbon Monoxide (CO) reading less than 5 parts per million (ppm) at Day 0.

Alcohol/Drugs.

* History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse.
* Current alcohol consumption that exceeds 25 standard drinks/week.
* Provide a breath alcohol concentration (BrAC) reading greater than .000 at Day 0.

Medical.

* Women who are pregnant, planning a pregnancy, and/or lactating.
* Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing the completion of procedures included within this protocol. Notable impairments will be evaluated by the Principal Investigator and eligibility will be determined on a case-by-case basis.
* Color blindness.
* Serious or unstable disease within the past 12 months (e.g. heart disease, cancer). Applicable conditions will be evaluated by the Principal Investigator and eligibility will be determined on a case-by-case basis.

Psychiatric.

* Lifetime history or current diagnosis of psychosis, bipolar disorder, and/or schizophrenia.
* Current diagnosis of major depression. Subjects with a history of major depression, in remission for 6 months or longer, are considered eligible.

Other.

* Any medical condition, extenuating circumstance, illness, disorder, adverse event (AE), and/or concomitant medication that could compromise participant safety and/or completion of the study procedures, as determined by the Principal Investigator. Subjects may be deemed ineligible or withdrawn for any of the aforementioned reasons at any point throughout the study.
* Non-compliance with the protocol and/or study design as determined by the Principal Investigator.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 316 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Daily Cigarette Rate (smoking behavior) | Days 0-50
  Daily cigarette consumption will be determined by the difference of unused cigarettes and used cigarette filters returned to the Center every Session after Day 0.The number of used cigarette filters and self-reported daily smoking rate will be recorded on a Smoking Rate Data Collection Form. We will examine changes in daily cigarette consumption averaged over each of the three 15-day pack periods.

SECONDARY OUTCOMES:
Smoking Topography | Days 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, & 50
  All lab cigarettes will be smoked using a smoking topography machine. This device is specifically designed to collect smoking topography variables. A cigarette is placed in a sterilized mouthpiece, and the internal pressure transducer measures pressure changes that occur during inhalation. The pressure changes are amplified, digitized and sampled at 1000 Hz, then software converts the signal to airflow (ml/s) in real time (s), and from this provides number of puffs, puff volume, puff duration, maximum flow, and interpuff interval (time between puffs). The primary topography outcome is total puff volume, due to its well- characterized responsiveness to changes in cigarette type. However, the smoking topography device collects additional measures that will be considered for exploratory analyses. The primary analyses to test study hypotheses will use average puff volume across clinic days within each period.
Subjective Cigarette Ratings | Days 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, & 50
  We will use our previous visual analog scale (VAS) to examine changes in subjective ratings using a 100 mm scale that has been used in previous smoking studies, including those used by the tobacco industry. Items include: strength, heat, draw, smoke smell, and burn rate. Composite ratings will be calculated in identical fashion to those described for the smoking topography outcome measures. Subjective cigarette ratings will be assessed after each cigarette smoked in the laboratory across all sessions.
Carbon Monoxide (CO) | Days 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, & 50
  CO measures will be assessed at the onset of each session, and then before and after each cigarette smoked in the lab. The device has a digital screen which reports CO in parts per million (ppm). Participants will provide a CO breath sample using standard procedures; the largest steady reading will be recorded as the recorded CO level.
Attitudes and Intentions (to use product) | Days 0, 5, 20, 35, & 50
  We will assess participants' attitudes and intentions toward the cigarette packs and their using the 'new' cigarette, similar to our previous work on cigarette smoking that applied the Reasoned Action Approach. We will use Likert-type semantic differential scales (likely to use/not use, using product is enjoyable/non enjoyable, harmful/not harmful). Because the study is designed to assess changes in smoking behavior and beliefs, the Theory of Reasoned Action would postulate that changes in product use would be mediated by changes in attitudes, and then intentions.
Cigarette Risk Beliefs | Days 0, 5, 20, 35, & 50
  To assess risk beliefs about participants' own brand of cigarettes on Day 0, we will use an 18-item, 5-point scale (1 = definitely not true; 5 = definitely true) including previously validated items assessing smokers' beliefs on cigarette harm. During applicable sessions post Day 0, participants will complete an 8-item, 5-point scale based on their assigned cigarettes. The Cigarette Risk Beliefs questionnaire will be administered on Day 0 before lab cigarette 1 (18-item baseline version), Day 5 before lab cigarette 1 and 2, Day 20 before lab cigarette 1 and 2, Day 35 before lab cigarette 1 and 2, and Day 50 before lab cigarette 1. The Cigarette Risk Beliefs questionnaire will be completed as the participant physically views a pack of their cigarette pack assignment (or own brand on Day 0) as per the randomization schema.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data and measures codebook will be made available after the conclusion of the study.

REFERENCES:
- [Derived] Stone MD, Mercincavage M, Wileyto EP, Tan ASL, Audrain-McGovern J, Villanti AC, Strasser AA. Effects of cigarette package colors and warning labels on marlboro smokers' risk beliefs, product appraisals, and smoking behavior: a randomized trial. BMC Public Health. 2023 Oct 27;23(1):2111. doi: 10.1186/s12889-023-17024-5. PMID 37891513
- [Derived] Mercincavage M, Albelda B, Mays D, Souprountchouk V, Giovenco DP, Audrain-McGovern J, Strasser AA. Shedding 'light' on cigarette pack design: colour differences in product perceptions, use and exposure following the US descriptor ban. Tob Control. 2022 Jan;31(1):19-24. doi: 10.1136/tobaccocontrol-2020-055886. Epub 2020 Sep 29. PMID 32994296